CLINICAL TRIAL: NCT07149857
Title: A Phase 2 Multicohort Trial to Further Characterize the Efficacy and Safety of Ciltacabtagene Autoleucel
Brief Title: A Study to Evaluate Efficacy and Safety of Ciltacabtagene Autoleucel
Acronym: CARTITUDE-10
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68284528MMY2012; 68284528MMY2012 (Other: Janssen Research & Development, LLC); 2025-521975-30-00 (Registry Identifier: EUCT number)
Expanded Access: Available
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Neoadjuvant Therapy; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants will undergo apheresis and continue to receive 1-2 more cycles of the induction regimen (DRd, VRd or DVRd regimen, in accordance with institution standard of care, and is not considered study treatment) that they were receiving prior to screening. After completion of induction therapy, participants will receive a conditioning regimen of cyclophosphamide daily for 3 days, followed by cilta-cel IV infusion on Day 1. Participants will later enter the post-treatment phase, which will start on Day 113 and last until end of study or cohort completion.
  Interventions: Drug: Cilta-cel; Drug: Cyclophosphamide; Drug: Induction therapy
- Cohort B (Experimental): Participants will undergo apheresis and continue to receive 1-2 more cycles of the induction regimen (DRd, VRd or DVRd regimen, in accordance with institution standard of care, and is not considered study treatment) that they were receiving prior to screening. After completion of induction therapy, participants will receive a conditioning regimen of cyclophosphamide and fludarabine daily for 3 days, followed by Ciltacel IV infusion on Day 1. Participants will later enter the post-treatment phase, which will start on Day 113 and last until end of study or cohort completion.
  Interventions: Drug: Cilta-cel; Drug: Cyclophosphamide; Drug: Induction therapy; Drug: Fludarabine

INTERVENTIONS:
Drug: Cilta-cel — Cilta-cel will be administered as intravenous infusion.
  Other Names: JNJ-68284528
Drug: Cyclophosphamide — Cyclophosphamide will be administered as intravenous infusion.
Drug: Induction therapy — Induction therapy consist of bortezomib, lenalidomide, and dexamethasone (VRd) or daratumumab, lenalidomide, and dexamethasone (DRd) or daratumumab, bortezomib, lenalidomide, and dexamethasone (DVRd), will will be administered.
Drug: Fludarabine — Fludarabine will be administered as intravenous infusion.
  Arms: Cohort B

SUMMARY:
The purpose of this study is to evaluate how well (efficacy) cilta-cel works when given with a fludarabine-free lymphodepletion regimen (a process of reducing the number of lymphocytes, a type of white blood cell in the body, typically through chemotherapy), or an alternative administration of cilta-cel infusion following a cyclophosphamide and fludarabine lymphodepletion regimen.

ELIGIBILITY:
Inclusion Criteria

* Documented diagnosis of newly diagnosed multiple myeloma (NDMM) according to the most recent international myeloma working group (IMWG) diagnostic criteria and measurable disease at diagnosis (prior to start of any anti-myeloma therapy): Serum monoclonal paraprotein (M-protein) level greater than equal to (>=)1.0 grams per deciliter (g/dL) or urine M-protein level >= 200 milligrams (mg)/24 hours; or light chain multiple myeloma in whom the only measurable disease is by serum free light chain (FLC) levels in the serum: involved serum free light chain >= 10 mg/dL and abnormal serum free light chain ratio
* Not considered a candidate for high-dose chemotherapy with stem cell transplantation due to: (a) Advanced age; or (b) Presence of comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with stem cell transplantation; or (c) Participant refusal of high-dose chemotherapy with stem cell transplantation as initial treatment
* Participant must have received at least 3 cycles and no more than 5 cycles of induction therapy. Initially, only participants receiving triplet induction therapy with DRd or VRd will be enrolled. Only after sponsor notification, participants receiving quadruplet DVRd induction therapy may be enrolled (screening can commence as early as during Cycle 3 of induction). Participants must have achieved >= partial response (PR) on the most recent disease assessment to be enrolled
* Eastern cooperative oncology group (ECOG) Performance Status score of 0 or 1
* Must be willing and able to adhere to the lifestyle restrictions specified in the protocol

Exclusion Criteria

* Frailty index of >= 2 according to Myeloma Geriatric Assessment score
* Known allergies, hypersensitivity, or intolerance to study intervention or its active agents
* Grade 2 or higher ongoing non-hematologic toxicity due to induction therapy, with the exception of grade 2 peripheral neuropathy due to bortezomib
* Participants who require continuous supplemental oxygen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-01-03 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD)-negative Complete Response (CR) After Cilta-cel Infusion | At least 12 months after Cilta-cel infusion on Day 1
  Participants in CR or better who achieve MRD-negative status at 12 months after cilta-cel infusion with a sensitivity of 10^-5, prior to progressive disease (PD) or subsequent anti-myeloma therapy will be reported.

SECONDARY OUTCOMES:
Overall MRD-negative CR Rate | From study start until progressive disease, subsequent therapy or end of study, whichever is earlier (Up to 3 years and 4 months)
  Overall MRD-negative CR is defined as the percentage of participants who achieve MRD-negative CR with a sensitivity of 10^-5 at any time after enrollment but prior to PD or subsequent anti-myeloma therapy.
CR or better status | From study start until progressive disease, subsequent therapy or end of study, whichever is earlier (Up to 3 years and 4 months)
  CR or better is defined as the percentage of participants who achieve a CR or stringent complete response (sCR) according to the most recent international myeloma working group (IMWG) criteria.
Progression Free Survival (PFS) | From study start until progressive disease, subsequent therapy or end of study, whichever is earlier (Up to 3 years and 4 months)
  PFS is defined as the time from the date of enrollment to the date of first documented PD, as defined in the most recent IMWG criteria, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 3 years and 4 months
  OS is measured from the date of enrollment to the date of the participant's death.
Number of Participants with Adverse Event (AE) by Severity | Up to 3 years and 4 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death related to adverse event.
Number of Participants with Abnormalities in Laboratory Parameters | Up to 3 years and 4 months
  Participants with abnormalities in laboratory parameters (hematology, chemistry) will be reported.
Levels of Cilta-cel T-Cell Expansion, and Persistence | Up to 3 years and 4 months
  Levels of Cilta-cel T cell expansion (proliferation), and persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.
Number of Participants with Anti-Cilta-Cel Antibodies | Up to 3 years and 4 months
  The presence of anti-cilta-cel antibodies will be determined from anti-drug antibody samples collected from each participant.
Percentage of Participants with Presence of Replication-competent Lentivirus (RCL) | Up to 3 years and 4 months
  Percentage of participants with presence of RCL will be reported.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown
  - Austin Hospital, Heidelberg
  - Fiona Stanley Hospital, Murdoch
- Spain (6):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency